CLINICAL TRIAL: NCT01892202
Title: Efficacy of C.E.R.A for Correction of Anemia and Maintenance of the Hb Levels in CKD Patients in Stage III - IV , Not on Dialysis , Treated According to Routine Clinical Practice
Brief Title: A Non-Interventional Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) in Patients With Chronic Kidney Disease Not on Dialysis
Status: No longer available | Type: Expanded Access
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25750
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Cohort Studies

INTERVENTIONS:
Other: Cohort

SUMMARY:
This multicenter observational study will evaluate the efficacy and safety of Mircera (methoxy polyethylene glycol-epoetin beta) in patients with chronic kidney disease not on dialysis in routine clinical practice. Eligible patients treated with Mircera for chronic renal anemia according to the standard of care and in line with the current local label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age inclusive
* Patients with chronic kidney disease Stage III-IV not on dialysis
* Hb < 10 g/dL (for correction of anemia) or Hb 10-12 g/dL and receiving any other ESA (for maintenance of Hb levels)
* Adequate iron status as judged by the treating physician

Exclusion Criteria:

* Hypersensitivity to recombinant human erythropoietin, polyethylene glycol or to any constituent of the study medication
* Significant acute or chronic bleeding
* Hemoglobinopathies (e.g. homozygous sickle-cell disease, thalassemia of all types)
* Active malignant disease during the last five years (except non-melanoma skin cancer)
* Uncontrolled or symptomatic secondary hyperparathyroidism
* Epileptic seizure during the last 6 months
* Poorly controlled hypertension (sitting blood pressure > 170/100 mmHG)
* Myocardial infarction or stroke, or severe or unstable CAD
* Severe liver disease during the previous 6 months
* Congestive heart failure NYHA Class III-IV
* Diagnosis or suspicion of pure red cell aplasia (PRCA)
* Planned elective surgery during the study period (except cataract surgery and vascular access surgery)
* Transfusion of red blood cells during the previous 2 months
* Pregnant women
* Any contra-indications to Mircera

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche